CLINICAL TRIAL: NCT04413552
Title: A Phase I, Double-blind, Placebo-controlled, Randomized, Single Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of INDV-2000 (C4X_3256) Under Fasting and Fed Conditions in Healthy Volunteers
Brief Title: INDV-2000 First in Human
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: INDV-2000-101; UG3DA050308 (NIH)
Record Dates: First submitted 2020-05-21; First posted 2020-06-04 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Part I - sequential escalating dose cohorts; within each dose cohort participants will be randomized to INDV-2000 or matching placebo in a 3:1 ratio.
  Part II - single cohort crossover study in which participants will receive INDV-2000 on 2 occasions separated by a 1-week washout period, once under fasting conditions and once after a standard high-fat breakfast.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part I: Double-blind;
  Part II: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part I: INDV-2000 (Experimental): Participants will receive a single dose of INDV-2000. The starting dose is 1 mg with dose escalation dependent upon observed clinical safety, tolerability and pharmacokinetics.
  Interventions: Drug: INDV-2000
- Part I: Placebo (Placebo Comparator): Participants will receive a single dose of matching placebo.
  Interventions: Drug: Placebo
- Part II: INDV-2000 Fasted/Fed (Experimental): Participants will receive a single dose of INDV-2000 orally on Day 1 under fasted conditions and a single dose of INDV-2000 after a high-fat breakfast on Day 8. Dose to be determined based on a well-tolerated dose studied in Part I.
  Interventions: Drug: INDV-2000

INTERVENTIONS:
Drug: INDV-2000 — INDV-2000 will be administered as either powder in solution or powder in capsule, depending on dose administered.
  Other Names: C4X_3256
  Arms: Part I: INDV-2000; Part II: INDV-2000 Fasted/Fed
Drug: Placebo — Placebo will be administered as either powder in solution or powder in capsule, depending on dose administered.
  Arms: Part I: Placebo

SUMMARY:
This study is a single ascending dose (SAD) study conducted to identify the maximum tolerated dose (MTD) of INDV-2000. After completion of the SAD portion of the study and acceptable safety evaluation, a food-interaction, single-dose study under fed and fasted conditions will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to verbalize understanding the consent form, able to provide written informed consent, and verbalize willingness to complete study procedures, and be able to comply with protocol requirements, rules and regulations of the study site, and be likely to complete all the study interventions.
* Must be considered a healthy male or non-childbearing female for Part I
* For Part II, must be a healthy male who did not participate in Part I and willing to consume a high-fat meal.
* Body mass index (BMI) within 18.0 to 30.0 kg/m^2, inclusive (minimum weight of at least 50.0 kg at Screening)
* Male subjects who are sexually active with female partners of child-bearing potential must use, with their partner, a condom plus an approved method of effective contraception from time of screening until 90 days after last dose of Investigational Medicinal Product (IMP). Additionally, male subjects must agree to not donate sperm during the study and for at least 90 days from last dose of IMP.

Exclusion Criteria:

* Have a medical history of clinically significant neurological, cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, or psychiatric disorder as judged by an Investigator,
* Have clinically significant abnormal biochemistry, hematology or urinalysis results as judged by an Investigator,
* Have a history of narcolepsy or other significant sleep disorders
* Have disorders that may interfere with drug absorption, distribution, metabolism and excretion (ADME) processes,
* Positive test results for human immunodeficiency virus (HIV)-1/HIV-2 antibodies, hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCVAb).
* Serious cardiac illness or other medical condition including, but not limited to: Uncontrolled arrhythmias; History of congestive heart failure (CHF); myocardial infarction < 6 months from receipt of first dose of IMP; uncontrolled symptomatic angina; corrected QT value (QTcF) > 450 msec for males and > 470 msec for females or history of prolonged QT syndrome; Have a blood pressure reading outside of the following range: systolic < 86 or > 149 mmHg; diastolic < 50 or > 94 mmHg
* Current active hepatic or biliary disease. Subjects with cholecystectomy < 90 days prior to screening.
* Regular alcohol consumption in males > 21 units per week and females > 14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine).
* Positive test result for alcohol and/or drugs of abuse at screening or prior to the first IMP administration.
* Current smokers and those who have smoked within the last 90 days. Current users of e-cigarettes and nicotine replacement products, and those who have used these products within the last 90 days.
* Concurrent treatment or treatment with an investigational drug within 30 days prior to the first dose.
* Blood donation of approximately 500 mL within 56 days or plasma donation within 7 days of screening.
* Subjects who are taking, or have taken, any prescribed or over-the-counter drugs (other than 2 g per day acetaminophen, hormone replacement therapy, hormonal contraception) or herbal remedies in the 14 days before IMP administration. Exceptions may apply on a case by case basis if considered not to interfere with the objectives of the study, as agreed by an Investigator and Sponsor's Medical Monitor.
* Any consumption of food or drink containing poppy seeds, grapefruit or Seville oranges within 7 days prior to the IMP administration
* Treatment with any known drugs that are moderate or strong inhibitors/inducers of cytochrome P450 (CYP) 3A4 within 30 days prior to first dose of IMP.
* Known allergy or hypersensitivity to IMP or its excipients.
* Any condition that, in the opinion of an Investigator, would interfere with evaluation of the IMP or interpretation of subject safety or study results.
* Affiliated with, or a family member of, site staff directly involved in the study, or anyone with a financial interest in the outcome of the study.
* Subjects who are unable, in the opinion of an Investigator, to comply fully with the study requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kankam, Principal Investigator — Altasciences Company Inc.
Locations (1):
- Altasciences Clinical Kansas, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers were enrolled at a single site in Overland Park, Kansas, United States.
Pre-assignment Details: This study was conducted in 2 parts: Part I was a double-blind, placebo-controlled, randomized, single ascending dose (SAD) study in which participants were randomized in cohorts of 8 subjects with 6 subjects receiving active drug and 2 subjects receiving placebo. Part II was an open-label, cross-over, food interaction, single-dose study with INDV-2000 administered once under fasting conditions and once after completion of a standard high-fat breakfast.
Groups:
- Part I: INDV-2000 1 mg: Participants received a single dose of 1 mg INDV-2000 orally under fasted conditions on Day 1.
- Part I: INDV-2000 5 mg: Participants received a single dose of 5 mg INDV-2000 orally under fasted conditions on Day 1.
- Part I: INDV-2000 20 mg: Participants received a single dose of 20 mg INDV-2000 orally under fasted conditions on Day 1.
- Part I: INDV-2000 50 mg: Participants received a single dose of 50 mg INDV-2000 orally under fasted conditions on Day 1.
- Part I: INDV-2000 120 mg: Participants received a single dose of 120 mg INDV-2000 orally under fasted conditions on Day 1.
- Part I: INDV-2000 180 mg: Participants received a single dose of 180 mg INDV-2000 orally under fasted conditions on Day 1.
- Part I: INDV-2000 360 mg: Participants received a single dose of 360 mg INDV-2000 orally under fasted conditions on Day 1.
- Part I: INDV-2000 720 mg: Participants received a single dose of 720 mg INDV-2000 orally under fasted conditions on Day 1.
- Part I: Pooled Placebo: Participants received a single dose of matching placebo orally under fasted conditions on Day 1.
- Part II: INDV-2000 360 mg Fasted/Fed: Participants received a single dose of 360 mg INDV-2000 orally on Day 1 under fasted conditions and a single dose of 360 mg INDV-2000 after a high-fat breakfast on Day 8.
Period: Overall Study
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg | Part I: Pooled Placebo | Part II: INDV-2000 360 mg Fasted/Fed
Started | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 6 | 16 | 8
Received Study Drug | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 8
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg | Part I: Pooled Placebo | Part II: INDV-2000 360 mg Fasted/Fed | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 8 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demographic data are reported separately for Part I and Part II.
  years
    Part I: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 0 | 64
    Part I | 42.0 (12.05) | 42.2 (12.80) | 34.3 (4.41) | 40.5 (10.93) | 33.5 (11.20) | 31.5 (12.36) | 44.3 (6.74) | 31.8 (11.34) | 36.5 (11.49) |  | 37.3 (11.02)
    Part II: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8
    Part II |  |  |  |  |  |  |  |  |  | 40.4 (7.52) | 40.4 (7.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 1 | 1 | 2 | 3 | 1 | 3 | 0 | 14
  Male | 5 | 4 | 6 | 5 | 5 | 4 | 3 | 5 | 13 | 8 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 6
  Not Hispanic or Latino | 6 | 6 | 5 | 6 | 4 | 5 | 6 | 5 | 15 | 8 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Black or African American | 1 | 3 | 4 | 2 | 0 | 2 | 3 | 4 | 9 | 4 | 32
  White | 5 | 2 | 1 | 4 | 4 | 4 | 3 | 2 | 7 | 4 | 36
  Other | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was considered related to study drug if it could not reasonably be explained by other factors.
  A serious AE is any event that met any of the following criteria:
  * Death
  * Life-threatening
  * In-patient hospitalization or prolongation of existing hospitalization
  * Persistent or significant disability/incapacity
  * Congenital anomaly/birth defect
  * Other important medical event that may have jeopardized the participant or required an intervention to prevent an above outcome.
  A severe AE describes the intensity of an AE, defined as causing marked limitation in activity; medical intervention or therapy or hospitalization required. For vital sign and laboratory abnormalities assessed as AEs, intensity was graded in accordance with the Food and Drug Administration Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, where Grade 3 = serious and Grade 4 = potentially life-threatening.
Time Frame: From first dose of study drug to end of study participation for each cohort; 11 days in Part 1 and 7 days in Part II, Period 1 (fasted conditions) and 10 days in Part II, Period 2 (fed conditions).
Population: Participants who received at least one dose of study drug (safety population)
Measure: Count of Participants; unit: Participants
Groups:
- Part I: INDV-2000 1 mg: Participants received a single dose of 1 mg INDV-2000 oral solution formulation under fasted conditions on Day 1.
- Part I: INDV-2000 5 mg: Participants received a single dose of 5 mg INDV-2000 oral solution formulation under fasted conditions on Day 1.
- Part I: INDV-2000 20 mg: Participants received a single dose of 20 mg INDV-2000 oral capsule formulation under fasted conditions on Day 1.
- Part I: INDV-2000 50 mg: Participants received a single dose of 50 mg INDV-2000 oral capsule formulation under fasted conditions on Day 1.
- Part I: INDV-2000 120 mg: Participants received a single dose of 120 mg INDV-2000 oral capsule formulation under fasted conditions on Day 1.
- Part I: INDV-2000 180 mg: Participants received a single dose of 180 mg INDV-2000 oral capsule formulation under fasted conditions on Day 1.
- Part I: INDV-2000 360 mg: Participants received a single dose of 360 mg INDV-2000 oral capsule formulation under fasted conditions on Day 1.
- Part I: INDV-2000 720 mg: Participants received a single dose of 720 mg INDV-2000 oral capsule formulation under fasted conditions on Day 1.
- Part II Period 1: INDV-2000 360 mg Fasted: Participants received a single dose of 360 mg INDV-2000 oral capsule formulation on Day 1 under fasted conditions.
- Part II Period 2: INDV-2000 360 mg Fed: Participants received a single dose of 360 mg INDV-2000 oral capsule formulation on Day 8 after a high-fat breakfast.
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg | Part I: Pooled Placebo | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 8 | 8
Participants
  Any treatment-emergent adverse event (TEAE) | 0 | 2 | 3 | 3 | 2 | 3 | 1 | 4 | 2 | 4 | 4
  Drug-related TEAE | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 4 | 0 | 4 | 3
  Treatment-emergent serious adverse events (TESAE) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Drug-related TESAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAE with grade 3 or higher toxicity | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  TEAE leading to discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatal TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Findings
Description: The investigator assessed abnormal laboratory values to determine clinical significance.
Time Frame: From first dose of study drug to end of study participation for each cohort; 11 days in Part I and 7 days in Part II, Period 1 (fasted conditions) and 10 days in Part II, Period 2 (fed conditions).
Population: Participants who received at least one dose of study drug (safety population)
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg | Part I: Pooled Placebo | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 8 | 8
Participants | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 1 | 2 | 0 | 0

3. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: The investigator assessed changes in vital signs (including including blood pressure, respiratory rate, heart rate and temperature) to determine clinical significance.
Time Frame: as for outcome 1
Population: Participants who received at least one dose of study drug (safety population)
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg | Part I: Pooled Placebo | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 8 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings
Description: The investigator assessed abnormal ECG values to determine clinical significance.
Time Frame: as for outcome 2
Population: Participants who received at least one dose of study drug (safety population)
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg | Part I: Pooled Placebo | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 8 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination Findings
Description: Any clinically significant abnormalities observed during physical examination, including changes from baseline, were recorded as adverse events on the adverse event (AE) case report form (CRF) and are reported in the adverse events section of results below. However, these events were not recorded as physical examination findings. Therefore, clinically significant physical examination findings can not be reported separately.
Time Frame: as for outcome 2
Population: Clinically significant physical examination findings were not recorded separately.
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg | Part I: Pooled Placebo | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Part I: Maximum Observed Plasma Concentration (Cmax) of INDV-2000 After a Single Dose
Description: Concentrations of INDV-2000 were measured using a validated high-performance liquid chromatography with electrospray tandem Mass spectrometry (LC-MS/MS) method. Pharmacokinetic parameters based on the actual sample collection times were derived using standard non-compartmental methods.
Time Frame: Day 1 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: Participants who received at least one dose of INDV-2000 and had an adequate number of pharmacokinetic (PK) samples collected to derive PK parameters (PK population).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 16.7 (3.93) | 87.6 (26.4) | 194 (33.3) | 489 (147) | 1000 (343) | 1100 (238) | 1880 (1140) | 2080 (688)

7. Secondary Outcome: Part I: Time to Maximum Observed Plasma Concentration (Tmax) of INDV-2000 After a Single Dose
Time Frame: Day 1 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: Participants who received at least one dose of INDV-2000 and had an adequate number of PK samples collected to derive PK parameters.
Measure: Median (Full Range); unit: hours
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 1.00 [0.58 to 2.08] | 0.50 [0.50 to 1.15] | 2.50 [1.00 to 3.05] | 2.02 [1.00 to 3.00] | 2.00 [1.00 to 2.00] | 3.50 [1.00 to 6.00] | 2.00 [2.00 to 3.00] | 3.00 [2.00 to 8.00]

8. Secondary Outcome: Part I: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUC0-last) of INDV-2000 After A Single Dose
Time Frame: Day 1 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng*h/mL | 67.3 (17.7) | 312 (181) | 915 (186) | 2340 (1020) | 6900 (4050) | 8520 (1600) | 17800 (9800) | 28700 (7810)

9. Secondary Outcome: Part I: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of INDV-2000 After A Single Dose
Time Frame: Day 1 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6
ng*h/mL | 69.5 (19.1) | 317 (180) | 907 (207) | 2350 (1030) | 6920 (4060) | 8530 (1590) | 17800 (9810) | 28700 (7810)

10. Secondary Outcome: Part I: Apparent Plasma Clearance (CL/F) of INDV-2000 After a Single Dose
Time Frame: Day 1 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: Participants who received at least one dose of INDV-2000 and had an adequate number of pharmacokinetic (PK) samples collected to derive PK parameters.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6
L/h | 15.4 (4.31) | 18.8 (6.98) | 23.2 (6.70) | 24.5 (9.67) | 22.4 (11.7) | 21.7 (4.03) | 25.8 (13.4) | 26.7 (7.78)

11. Secondary Outcome: Part I: Plasma Terminal Half-life of INDV-2000 After a Single Dose
Time Frame: Day 1 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6
hours | 2.19 (0.32) | 2.52 (0.46) | 2.56 (0.37) | 2.81 (0.47) | 3.56 (1.18) | 3.47 (0.46) | 4.57 (0.58) | 5.28 (2.18)

12. Secondary Outcome: Part I: Maximum Observed Plasma Concentration (Cmax) of M12 After a Single Dose of INDV-2000
Description: Concentrations of INDV-2000 metabolite M12 were measured using a validated high-performance liquid chromatography with electrospray tandem Mass spectrometry (LC-MS/MS) method.
Time Frame: Day 1 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 12.2 (3.31) | 76.4 (14.4) | 182 (34.0) | 372 (113) | 983 (121) | 963 (326) | 1650 (536) | 1840 (318)

13. Secondary Outcome: Part I: Time to Maximum Observed Plasma Concentration (Tmax) of M12 After a Single Dose of INDV-2000
Time Frame: Day 1 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 1.08 [1.00 to 2.08] | 0.50 [0.50 to 1.15] | 3.50 [1.00 to 4.00] | 2.52 [1.00 to 4.00] | 3.00 [3.00 to 4.00] | 4.00 [4.00 to 6.00] | 3.00 [2.00 to 8.00] | 3.00 [3.00 to 8.00]

14. Secondary Outcome: Part I: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration of M12 After A Single Dose of INDV-2000
Time Frame: Day 1 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng*h/mL | 72.8 (28.8) | 413 (223) | 1300 (489) | 3190 (2250) | 10000 (4370) | 10100 (5540) | 24000 (16200) | 25800 (6120)

15. Secondary Outcome: Part I: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of M12 After A Single Dose of INDV-2000
Time Frame: Day 1 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng*h/mL | 74.8 (30.3) | 417 (222) | 1310 (489) | 3200 (2240) | 10100 (4370) | 10100 (5540) | 24000 (16200) | 25800 (6110)

16. Secondary Outcome: Part I: Plasma Terminal Half-life of M12 After a Single Dose of INDV-2000
Time Frame: Day 1 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 3.78 (0.84) | 4.04 (0.73) | 3.93 (0.50) | 4.23 (1.21) | 4.51 (0.81) | 4.45 (0.56) | 5.54 (1.07) | 5.87 (2.08)

17. Secondary Outcome: Part II: Cmax of INDV-2000 After a Single Dose Under Fasting and Fed Conditions
Time Frame: Day 1 and Day 8 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: The food effect PK population included the subset of Part II participants in the PK population who had at least one evaluable PK parameter for at least one meal condition.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
Number analyzed (Participants) | 8 | 8
ng/mL | 1700 (584) | 2720 (796)

18. Secondary Outcome: Part II: Tmax of INDV-2000 After a Single Dose Under Fasting and Fed Conditions
Time Frame: Day 1 and Day 8 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
Number analyzed (Participants) | 8 | 8
hours | 3.00 [2.00 to 6.00] | 3.00 [1.00 to 4.00]

19. Secondary Outcome: Part II: AUC0-last of INDV-2000 After a Single Dose Under Fasting and Fed Conditions
Time Frame: Day 1 and Day 8 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
Number analyzed (Participants) | 8 | 8
ng*hr/mL | 18200 (6060) | 16700 (7970)

20. Secondary Outcome: Part II: AUC0-inf of INDV-2000 After a Single Dose Under Fasting and Fed Conditions
Time Frame: Day 1 and Day 8 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
Number analyzed (Participants) | 6 | 8
ng*hr/mL | 19700 (7690) | 17400 (8130)

21. Secondary Outcome: Part II: Apparent Clearance of INDV-2000 After a Single Dose Under Fasting and Fed Conditions
Time Frame: Day 1 and Day 8 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
Number analyzed (Participants) | 6 | 8
L/hr | 21.2 (9.61) | 24.1 (9.04)

22. Secondary Outcome: Part II: Plasma Terminal Half-life of INDV-2000 After a Single Dose Under Fasting and Fed Conditions
Time Frame: Day 1 and Day 8 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
Number analyzed (Participants) | 6 | 8
hours | 6.37 (1.62) | 2.91 (0.76)

23. Secondary Outcome: Part II: Cmax of M12 After a Single Dose of INDV-2000 Under Fasting and Fed Conditions
Time Frame: Day 1 and Day 8 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
Number analyzed (Participants) | 8 | 8
ng/mL | 1320 (243) | 1500 (277)

24. Secondary Outcome: Part II: Tmax of M12 After a Single Dose of INDV-2000 Under Fasting and Fed Conditions
Time Frame: Day 1 and Day 8 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
Number analyzed (Participants) | 8 | 8
hours | 4.00 [2.00 to 6.00] | 4.00 [2.00 to 8.00]

25. Secondary Outcome: Part II: AUC0-last of M12 After a Single Dose of INDV-2000 Under Fasting and Fed Conditions
Time Frame: Day 1 and Day 8 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
Number analyzed (Participants) | 8 | 8
ng*hr/mL | 15800 (4180) | 15000 (3920)

26. Secondary Outcome: Part II: AUC0-inf of M12 After a Single Dose of INDV-2000 Under Fasting and Fed Conditions
Time Frame: Day 1 and Day 8 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
Number analyzed (Participants) | 7 | 8
ng*hr/mL | 18200 (4030) | 15800 (4300)

27. Secondary Outcome: Part II: Plasma Terminal Half-life of M12 After a Single Dose of INDV-2000 Under Fasting and Fed Conditions
Time Frame: Day 1 and Day 8 pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
Number analyzed (Participants) | 7 | 8
hours | 7.43 (1.13) | 5.21 (1.24)

ADVERSE EVENTS:
Time Frame: From first dose of study drug to end of study participation for each cohort; 11 days in Part 1 and 7 days in Part II, Period 1 (fasted conditions) and 10 days in Part II, Period 2 (fed conditions).
Description: All-cause mortality is reported for all randomized (in Part I) and enrolled (Part II) participants. Adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Part I: INDV-2000 1 mg | Part I: INDV-2000 5 mg | Part I: INDV-2000 20 mg | Part I: INDV-2000 50 mg | Part I: INDV-2000 120 mg | Part I: INDV-2000 180 mg | Part I: INDV-2000 360 mg | Part I: INDV-2000 720 mg | Part I: Pooled Placebo | Part II Period 1: INDV-2000 360 mg Fasted | Part II Period 2: INDV-2000 360 mg Fed
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/16 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/16 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6 | 3/6 | 3/6 | 2/6 | 3/6 | 1/6 | 4/6 | 2/16 | 4/8 | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: INDV-2000 1 mg (N=6) | Part I: INDV-2000 5 mg (N=6) | Part I: INDV-2000 20 mg (N=6) | Part I: INDV-2000 50 mg (N=6) | Part I: INDV-2000 120 mg (N=6) | Part I: INDV-2000 180 mg (N=6) | Part I: INDV-2000 360 mg (N=6) | Part I: INDV-2000 720 mg (N=6) | Part I: Pooled Placebo (N=16) | Part II Period 1: INDV-2000 360 mg Fasted (N=8) | Part II Period 2: INDV-2000 360 mg Fed (N=8)
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 0 | 4 | 3
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure diastolic increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI will not disseminate, present or publish any of the study data without the prior written approval from Indivior to do so.

DOCUMENTS (3):
  • Study Protocol (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT04413552/Prot_001.pdf
  • Statistical Analysis Plan (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT04413552/SAP_002.pdf
  • Informed Consent Form (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT04413552/ICF_000.pdf